CLINICAL TRIAL: NCT01233557
Title: Measurement of Biomarkers of Bone Resorption in Patients With Hormone Sensitive Bone Metastases From Prostate Cancer Treated With Antiandrogen Therapy and Bisphosphonates
Brief Title: Biomarkers of Bone Resorption in Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 10/S0802/36
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bone Metastases

SUMMARY:
Biomarkers of bone resorption will be measured in the blood of patients with bone metastases from prostate cancer during the course of their illness. Changes in these biomarkers will be correlated with the patient's treatment with antiandrogen therapy and bisphosphonates and the response and/or progression of their cancer. It is hoped that serial measurement of these biomarkers may allow therapeutic monitoring in the future with successful individualisation of bisphosphonate therapy for metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer with bone metastases
* hormone sensitive

Exclusion Criteria:

* inadequate renal function
* ongoing dental problems
* previous bisphosphonate therapy

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men with hormone sensitive prostate cancer with bone metastases
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Bissett, M.D., Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom